CLINICAL TRIAL: NCT06461845
Title: Effect of Whole Body Vibration Effect on Trunk Control, Functional Performance and Selective Control of Lower Extremity in Children With Cerebral Palsy
Brief Title: Whole Body Vibration Effect on Trunk Control, Functional Performance and Selective Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/PCR&AHS/23/0771
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy
Keywords: Whole body vibration; cerebral palsy; trunk control; muscle performance; selective motor control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration group (Experimental)
  Interventions: Other: Whole Body Vibration group; Other: conventional therapy
- conventional therapy group (Active Comparator)
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Whole Body Vibration group — This group will be given WBV training session, by using a WBV platform was conducted to the study group. The wBV program comprises various positions such as the child stands in an erect position, sitting, and in kneeling position on vibrating platform. This platform vibrates horizontally at a frequency ranged from 10 to 25 Hz. The participants had to carry out each position for 2 min in the first month, and then it was increased to 3 min in the second month. The rest period between each position was 1 min in the first month, then it became half a minute in the second month. The duration of the vibration exposure was 10 min.
  Arms: whole body vibration group
Other: conventional therapy — This group will be provided with the conventional physical therapy. To this, stretching activities to keep up muscle elasticity particularly Achilles tendon, hamstring muscles, hip flexors and adductors; strength training to hip flexor, knee extensor, and ankle dorsiflexor;

SUMMARY:
Permanent neurological disorders such as cerebral palsy lead to problems with motor, sensory, and cognitive functions, which in turn limit one's ability to do certain activities. While the exact causes of cerebral palsy differ from child to child, anoxia-induced brain injury is a major cause of the disorder. The body parts affected, tone, and involuntary motions are used to categorise cerebral palsy. Among all the forms, spastic CP is the most prevalent. In individuals with CP, postural stabilisation and adaptations of the head, trunk, pelvic, and shoulder girdles grow more slowly. The primary problem with CP children is their gross movement pattern, which prevents them from performing single joint movements. Muscle strength increases significantly with WBV exercise training, which also reduces spasticity and enhances CP children's motor function. This study is important because it will determine whether WBV improves trunk control, functional performance, and lower limb selective control.

Data from Rising Sun Institute will be gathered for this randomised clinical trial. 38 patients will be included in the study. The study's inclusion criteria will include CP children with ages between 6 and 12 years old, those who can stand or walk alone (even with unusual gait patterns), GMFCS I and II, and children with diplegic cerebral palsy. Children with cerebral palsy (CP) who have had a lower limb fracture, fixed contracture, or other deformity, as well as those who have had a botulinum toxin injection or selective dorsal rhizotomy within the last six months, will not be eligible. Stretching exercises, strengthening exercises, trunk control facilitation, and rightening reaction facilitation will be the specific physical therapy treatments administered to group A. In addition, group B will receive WBV in addition to the specific physical therapy treatments (stretching exercises, strengthening exercises, trunk control facilitation, and rightening reaction facilitation). For two months, the 30-minute sessions will be held three times a week. The Modified Trost Test will test selective lower limb control, the PEDI scale will assess functional performance, and the Trunk Control Measurement Scale will monitor trunk stability before and after sessions. SPSS version 26 will be utilised for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Childrens who follow verbal command

  * Childrens who can stand or walk alone (either with altered pattern)
  * Age limit: 6 -12 years
  * GMFCS I & II
  * Diplegic Cerebral palsy

Exclusion Criteria:

* • Childrens with history of fracture in last 6 months

  * Childrens with fixed contracture or other deformity of lower limb
  * Childrens having visual or auditory impairments
  * Selective dorsal rhizotomy or botulinum toxin injection to lower extremities within past six months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
.Trunk Control Measurement Scale (TCMS) for trunk control | Baseline to 8 weeks
  To access trunk control in CP child we choose TCMS, it assesses seated trunk control in three dimensions static sitting balance, dynamic sitting balance and dynamic reaching. The maximum score is 58 points. The items are scored from 0 to 3, with 0 being the inability to perform the task and 3 being the complete performance of the item (20).
Modified Trost Test for selective control of lower extremity | Baseline to 8 weeks
  This test is used for assessment of selective motor control of lower extremity. It is a 3-point scale with assessment of ankle dorsiflexion, knee extension, hip flexion and hip abduction.
  * 0 point for Only patterned movement observed (total synergy)
  * 1 for Partially isolated movement observed (partial synergy)
  * 2 for Completely isolated movement observed (no synergy)
PEDI SCALE for functional performance | Baseline to 8 weeks
  This scale is use for assessment of functional performance. It is composed of 197 items, subdivided into three domains(22).
  Mobility (59 items, involving tub transfers, toilet transfers, indoor and outdoor locomotion, and climbing stairs); Self-care (73 items involving eating, dressing, grooming); Social function (65 items related to communication with comprehension and expression, problem-solving, interactions with peers and adults and safety awareness).
  Each item scores (0) for "unable" to perform the activities or (1) for "capable

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Society for Rehabilitation of Disabled, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annino G, Alashram AR, Alghwiri AA, Romagnoli C, Messina G, Tancredi V, Padua E, Mercuri NB. Effect of segmental muscle vibration on upper extremity functional ability poststroke: A randomized controlled trial. Medicine (Baltimore). 2019 Feb;98(7):e14444. doi: 10.1097/MD.0000000000014444. PMID 30762754
- [Background] Ali YMM, Elhadidy EI, Abdou RGE, Darwish SY. EFFECT OF WHOLE BODY VIBRATION ON QUADRICEPS MUSCLE PERFORMANCE IN HEMIPARETIC CHILDREN. 11. Ahmadizadeh Z, Khalili MA, Ghalam MS, Mokhlesin M. Effect of whole body vibration with stretching exercise on active and passive range of motion in lower extremities in children with cerebral palsy: A randomized clinical trial. Iranian Journal of Pediatrics. 2019;29(5)
- [Background] Telford D, Vesey RM, Hofman PL, Gusso S. The Effect of Vibration Therapy on Walking Endurance in Children and Young People With Cerebral Palsy: Do Age and Gross Motor Function Classification System Matter? Arch Rehabil Res Clin Transl. 2020 Jun 20;2(3):100068. doi: 10.1016/j.arrct.2020.100068. eCollection 2020 Sep. PMID 33543094